CLINICAL TRIAL: NCT01187407
Title: A Randomized, Placebo-Controlled, Double-Blind Study of LY2216684 Flexible-Dose 12 mg to 18 mg Once Daily and LY2216684 Fixed-Dose 6 mg Once Daily as Adjunctive Treatment for Patients With Major Depressive Disorder Who Are Partial Responders to Selective Serotonin Reuptake Inhibitor Treatment
Brief Title: A Study of Flexible or Fixed Dose LY2216684 as Adjunctive Treatment for Participants With Major Depressive Disorder Who Have Had a Partial Response to Selective Serotonin Reuptake Inhibitor (SSRI) Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12182; H9P-MC-LNBQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-08-20; First posted 2010-08-24 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 12 or 18 mg flexible dose LY2216684 + SSRI (Experimental): LY2216684: flexible dose of 12 or 18 milligrams (mg), administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Prior to entering the Adjunctive Treatment (AT) Phase, participants completed a 3-week Confirmation (CF) Phase where they received placebo (orally, QD) adjunctive to their SSRI. After the CF Phase, and after randomization criteria were met, participants were randomized to a 12 or 18 mg flexible dose of LY2216684.
  During the AT Phase, participants first received 6 mg LY2216684 QD for 3 days, followed by 12 mg QD for the next 11 days. Then, based on efficacy and tolerability, dosage could be increased to 18 mg QD over the next 6 weeks. Participants on 18 mg QD could have had their dose decreased back to 12 mg QD. Participants who completed the AT Phase or discontinued early had the option to enter the Discontinuation (DC) Phase.
  During the 1-week abrupt DC Phase, participants maintained their SSRI treatment.
  Interventions: Drug: LY2216684; Drug: Placebo; Drug: SSRI
- 6 mg fixed dose LY2216684 + SSRI (Experimental): LY2216684: fixed dose of 6 mg, administered orally, QD for 8 weeks, adjunctive to an SSRI
  Prior to entering the AT Phase, participants completed a 3-week CF Phase where they received placebo (orally, QD) adjunctive to their SSRI. After the CF Phase, and after randomization criteria were met, participants were randomized to 6 mg fixed dose of LY2216684.
  During the AT Phase, participants received a 6 mg fixed dose of LY2216684 adjunctive to their SSRI for 8 weeks. Participants who completed the AT Phase or discontinued early had the option to enter the DC Phase.
  During the 1-week abrupt DC Phase, participants maintained their SSRI treatment.
  Interventions: Drug: LY2216684; Drug: Placebo; Drug: SSRI
- Placebo + SSRI (Placebo Comparator): Placebo: administered orally, QD for 8 weeks, adjunctive to an SSRI
  Prior to entering the AT Phase, participants completed a 3-week CF Phase where they received placebo (orally, QD) adjunctive to their SSRI. After the CF Phase, and after randomization criteria were met, participants were randomized to placebo.
  During the AT Phase, participants received placebo (administered orally, QD) adjunctive to their SSRI for 8 weeks. Participants who completed the AT Phase or discontinued early had the option to enter the DC Phase.
  During the 1-week abrupt DC Phase, participants maintained their SSRI treatment.
  Interventions: Drug: Placebo; Drug: SSRI

INTERVENTIONS:
Drug: LY2216684
  Other Names: Edivoxetine
  Arms: 12 or 18 mg flexible dose LY2216684 + SSRI; 6 mg fixed dose LY2216684 + SSRI
Drug: Placebo
Drug: SSRI — Participants should have been on their SSRI for at least 6 weeks prior and were to continue on their stable dose throughout the study
  Other Names: selective serotonin reuptake inhibitor

SUMMARY:
The purpose of this study is to assess if LY2216684 (flexible dose of 12 to 18 milligrams [mg] or fixed dose of 6 mg once daily) is superior to placebo once daily in the adjunctive treatment of participants with Major Depressive Disorder (MDD) who were identified as partial responders to an adequate course of treatment with a selective serotonin reuptake inhibitor (SSRI) during an 8-week, double-blind, acute adjunctive treatment phase.

DETAILED DESCRIPTION:
Following the Confirmation (CF) Phase, participants were randomized to adjunctive LY2216684 or adjunctive placebo if they had <25% improvement in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score over the past 3 weeks and a current MADRS total score ≥14. Participants who did not meet criteria received adjunctive placebo to preserve the blind.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Major Depressive Disorder (MDD)
* Using a reliable method of birth control
* Are taking a selective serotonin reuptake inhibitor (SSRI) approved for MDD treatment within the participant's country and the SSRI prescribed, including dose, should be consistent with labeling guidelines within the participating country
* Have a partial response to SSRI treatment
* Meet inclusion scores on pre-defined psychiatric scales to assess diagnosis of depression, disease severity, and response to SSRI treatment
* Reliable and able to keep all scheduled appointments

Exclusion Criteria:

* Presence of another primary psychiatric illness:

  * Have had or currently have any additional ongoing Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) Axis 1 condition other than major depression within 1 year of screening
  * Have had any anxiety disorder that was considered a primary diagnosis within the past year (including panic disorder, obsessive-compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder, and social phobia, but excluding specific phobias)
  * Have a current or previous diagnosis of a bipolar disorder, schizophrenia, or other psychotic disorder
  * Have a history of substance abuse and/or dependence within the past 1 year (drug categories defined by DSM-IV-TR), not including caffeine and nicotine
  * Have an Axis II disorder that, in the judgment of the investigator, would interfere with compliance with protocol
* Have any diagnosed medical condition that could be exacerbated by noradrenergic agents, including unstable hypertension, unstable heart disease, tachycardia, tachyarrhythmia, narrow-angle glaucoma, and history of urinary hesitation or retention
* Use of excluded concomitant or psychotropic medication other than SSRI
* Have initiated or discontinued hormone therapy within the previous 3 months of prior to enrollment
* History of treatment-resistant depression as shown by lack of response of the current depressive episode to 2 or more adequate courses of antidepressant therapy at a clinically appropriate dose for at least 4 weeks, or in the judgment of the investigator, the participant has treatment-resistant depression
* Have a lifetime history of vagal nerve stimulation (VNS) transcranial magnetic stimulation (TMS), or psychosurgery
* Have received electroconvulsive therapy (ECT) in the past year
* Enrollment in a clinical study for an investigational drug
* Serious or unstable medical condition
* History of seizure disorders
* Have initiated psychotherapy, change in intensity of psychotherapy or other nondrug therapies (such as acupuncture or hypnosis) within 6 weeks prior to enrollment or any time during the study
* Participants who, in the opinion of the investigator, are judged to be at serious risk for harm to self or others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1480 (Actual)
Dates: Start 2011-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (54):
- United States (28):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chino, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Imperial, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., National City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherman Oaks, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colorado Springs, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clearwater, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coral Gables, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoffman Estates, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haverhill, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Weymouth, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flowood, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., O'Fallon, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
- Croatia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rab
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- Czechia (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hořovice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hostivice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kladno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olomouc
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strakonice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ústí nad Labem
- Finland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsinki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Joensuu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuopio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampere
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Turku
- Japan (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico
- Slovakia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Košice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Michalovce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rimavská Sobota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rožňava

REFERENCES:
- [Derived] Stauffer VL, Liu P, Goldberger C, Marangell LB, Nelson C, Gorwood P, Fava M. Is the Noradrenergic Symptom Cluster a Valid Construct in Adjunctive Treatment of Major Depressive Disorder? J Clin Psychiatry. 2017 Mar;78(3):317-323. doi: 10.4088/JCP.15m09972. PMID 27685842
- [Derived] Ball SG, Ferguson MB, Martinez JM, Pangallo BA, Nery ES, Dellva MA, Sparks J, Zhang Q, Liu P, Bangs M, Goldberger C. Efficacy outcomes from 3 clinical trials of edivoxetine as adjunctive treatment for patients with major depressive disorder who are partial responders to selective serotonin reuptake inhibitor treatment. J Clin Psychiatry. 2016 May;77(5):635-42. doi: 10.4088/JCP.14m09619. PMID 27035159

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The first 3 weeks of the study was a double-blind Confirmation Phase during which participants continued to receive their SSRI with adjunctive placebo. If randomization criteria were met, participants were randomized to adjunctive LY2216684 or adjunctive placebo. If criteria were not met, participants continued on placebo to maintain the blind.
Groups:
- Placebo + SSRI (Pre-randomized Participants): Placebo: administered orally, once daily (QD) for 3 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
- 12 or 18 mg LY2216684 + SSRI (Randomized Participants): LY2216684: flexible dose of 12 or 18 milligrams (mg), administered orally, QD for 8 weeks, adjunctive to an SSRI
- 6 mg LY2216684 + SSRI (Randomized Participants): LY2216684: fixed dose of 6 mg, administered orally, QD for 8 weeks, adjunctive to an SSRI
- Placebo + SSRI (Randomized Participants); Placebo + SSRI (Non-randomized Participants): Placebo: administered orally, QD for 8 weeks, adjunctive to an SSRI
Period: Confirmation (CF) Phase, 3 Weeks
Arm/Group | Placebo + SSRI (Pre-randomized Participants) | 12 or 18 mg LY2216684 + SSRI (Randomized Participants) | 6 mg LY2216684 + SSRI (Randomized Participants) | Placebo + SSRI (Randomized Participants) | Placebo + SSRI (Non-randomized Participants)
Started | 1480 | 0 | 0 | 0 | 0
Entered Discontinuation (DC) Phase | 25 (Participants who discontinued the CF Phase early had the option to enter the DC Phase.) | 0 | 0 | 0 | 0
Completed | 1390 (Participants who completed the CF Phase entered the Adjunctive Treatment (AT) Phase.) | 0 | 0 | 0 | 0
Not Completed | 90 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 29 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 13 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 29 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 4 | 0 | 0 | 0 | 0
Period: Adjunctive Treatment (AT) Phase, 8 Weeks
Arm/Group | Placebo + SSRI (Pre-randomized Participants) | 12 or 18 mg LY2216684 + SSRI (Randomized Participants) | 6 mg LY2216684 + SSRI (Randomized Participants) | Placebo + SSRI (Randomized Participants) | Placebo + SSRI (Non-randomized Participants)
Started | 0 | 232 | 226 | 231 | 701
Entered Discontinuation (DC) Phase | 0 | 212 (Participants who completed the AT Phase or discontinued early had the option to enter the DC Phase.) | 215 (Participants who completed the AT Phase or discontinued early had the option to enter the DC Phase.) | 220 (Participants who completed the AT Phase or discontinued early had the option to enter the DC Phase.) | 660 (Participants who completed the AT Phase or discontinued early had the option to enter the DC Phase.)
Completed | 0 | 196 | 191 | 202 | 626
Not Completed | 0 | 36 | 35 | 29 | 75
Not completed — Adverse Event | 0 | 13 | 6 | 5 | 12
Not completed — Lack of Efficacy | 0 | 3 | 8 | 5 | 13
Not completed — Lost to Follow-up | 0 | 3 | 5 | 2 | 9
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 6 | 5 | 3 | 10
Not completed — Withdrawal by Subject | 0 | 9 | 9 | 11 | 22
Not completed — Sponsor Decision | 0 | 2 | 2 | 2 | 7

BASELINE CHARACTERISTICS:
Population: Participants who completed the Confirmation (CF) Phase and were randomized to adjunctive LY2216684 or adjunctive placebo or who did not meet randomization criteria and continued on placebo to maintain the blind.
Groups:
- 12 or 18 mg LY2216684 + SSRI (Randomized Participants): LY2216684: flexible dose of 12 or 18 milligrams (mg), administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
- Total: Total of all reporting groups
Arm/Group | 12 or 18 mg LY2216684 + SSRI (Randomized Participants) | 6 mg LY2216684 + SSRI (Randomized Participants) | Placebo + SSRI (Randomized Participants) | Placebo + SSRI (Non-randomized Participants) | Total
Number analyzed (Participants) | 232 | 226 | 231 | 701 | 1390
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.63 (12.00) | 47.06 (12.76) | 47.30 (12.10) | 46.35 (12.42) | 46.67 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 153 | 156 | 465 | 923
  Male | 83 | 73 | 75 | 236 | 467
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 14 | 49 | 83
  Not Hispanic or Latino | 183 | 181 | 178 | 562 | 1104
  Unknown or Not Reported | 38 | 36 | 39 | 90 | 203
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 3 | 4 | 8
  Asian | 21 | 26 | 20 | 54 | 121
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 16 | 25 | 18 | 63 | 122
  White | 192 | 173 | 186 | 572 | 1123
  More than one race | 2 | 2 | 3 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 103 | 98 | 104 | 377 | 682
  Czechia | 44 | 44 | 46 | 119 | 253
  Slovakia | 33 | 35 | 34 | 39 | 141
  Finland | 18 | 12 | 17 | 61 | 108
  Croatia | 9 | 10 | 7 | 26 | 52
  Japan | 20 | 23 | 19 | 53 | 115
  Hungary | 2 | 2 | 1 | 3 | 8
  Romania | 3 | 2 | 3 | 23 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Randomization to Week 8 in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist (sadness [apparent], sadness [reported], inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts). Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: All randomized participants who have non-missing values at the time of randomization and at least one post-randomization value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- 12 or 18 mg Flexible Dose LY2216684 + SSRI: LY2216684: flexible dose of 12 or 18 milligrams (mg), administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
- 6 mg Fixed Dose LY2216684 + SSRI: LY2216684: fixed dose of 6 mg, administered orally, QD for 8 weeks, adjunctive to an SSRI
- Placebo + SSRI: Placebo: administered orally, QD for 8 weeks, adjunctive to an SSRI
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 231 | 220 | 228
units on a scale | -9.36 (0.55) | -9.59 (0.55) | -9.36 (0.54)
Statistical Analysis 1: Comparison: 12 or 18 mg Flexible Dose LY2216684 + SSRI vs Placebo + SSRI; Test type: Superiority or Other; p = 0.997, Mixed Models Analysis — Primary comparison
Statistical Analysis 2: Comparison: 6 mg Fixed Dose LY2216684 + SSRI vs Placebo + SSRI; Test type: Superiority or Other; p = 0.769, Mixed Models Analysis — Secondary comparison

2. Secondary Outcome: Change From Randomization to Week 8 in the Sheehan Disability Scale (SDS) Global Functional Impairment Score
Description: The SDS was completed by the participant and used to assess the effect of the participant's symptoms on their work (Item 1), social (Item 2), and family life (Item 3). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. The Global Functional Impairment Score is the sum of the 3 items, and scores ranged from 0 to 30 with higher values indicating greater disruption in the participant's work life (work/school impairment score), social life (social life/leisure activities impairment score), and family life (family life/home responsibilities impairment score). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 225 | 210 | 221
units on a scale | -5.30 (0.43) | -6.29 (0.44) | -4.30 (0.43)

3. Secondary Outcome: Change From Randomization to Week 8 in the Fatigue Associated With Depression (FAsD) Impact Subscale Score
Description: The FAsD is a participant-rated scale with a total of 13 items. Six of the 13 items ask how often participants experience different aspects of fatigue with responses from 1 (never) to 5 (always). Seven of the 13 items ask how often fatigue impacts various aspects of the participant's lives with responses from 1 (not at all) to 5 (very much). The impact subscale score was derived by taking the mean of Items 7 through 13 (applicable items only). Item 12 applied only to participants with a spouse or significant other and Item 13 applied to participants who had a job or who went to school. The FAsD impact subscale score ranges from 1 to 5. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline subscale score, treatment-by-visit, and baseline subscale score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 225 | 210 | 221
units on a scale | -0.71 (0.06) | -0.67 (0.06) | -0.56 (0.06)

4. Secondary Outcome: Percentage of Participants Achieving a Montgomery-Asberg Depression Rating Scale (MADRS) Total Score of Less Than or Equal to 10 up to Week 8
Description: A MADRS total score of less than or equal to 10 was defined as remission criteria. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist (sadness [apparent], sadness [reported], inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts). Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Percentage of participants was calculated by dividing the number of participants who meet criteria for remission by the total number of participants analyzed, multiplied by 100%.
Time Frame: Randomization up to 8 weeks
Population: All randomized participants who have non-missing values at the time of randomization and at least one post-randomization value. Last observation carried forward (LOCF) methodology was used.
Measure: Number; unit: percentage of participants
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 231 | 221 | 228
percentage of participants | 26.84 | 29.41 | 26.32

5. Secondary Outcome: Percentage of Participants Achieving a Montgomery-Asberg Depression Rating Scale (MADRS) Total Score of Less Than or Equal 10 for at Least 2 Consecutive Measurements, Including the Participant's Last Measurement
Description: A MADRS total score of less than or equal to 10 for at least 2 consecutive measurements, including the participant's last measurement was defined as remission criteria at last 2 consecutive visits. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist (sadness [apparent], sadness [reported], inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts). Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Percentage of participants was calculated by dividing the number of participants who meet criteria for remission at last 2 consecutive visits by the total number of participants analyzed, multiplied by 100%.
Time Frame: Randomization up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 231 | 221 | 228
percentage of participants | 17.75 | 19.00 | 14.47

6. Secondary Outcome: Change From Randomization to Week 8 in the Hospital and Anxiety and Depression Scale (HADS) Anxiety Subscale Score
Description: The HADS is a 14-item questionnaire with 2 subscales: anxiety and depression. Each item was rated on a 4-point scale (0 to 3), giving maximum scores of 21 for anxiety and depression subscale. Scores of 11 or more on either subscale were considered to be a significant 'case' of psychological morbidity, while scores of 8 to 10 represent 'borderline' and scores of 0 to 7 represent 'normal'. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline subscale score, treatment-by-visit, and baseline subscale score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 231 | 220 | 228
units on a scale | -2.24 (0.24) | -2.64 (0.24) | -2.05 (0.24)

7. Secondary Outcome: Percentage of Participants Who Have a Greater Than or Equal to 50 Percent Improvement in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Randomization up to Week 8
Description: A greater than or equal to 50 percent improvement (that is, a decrease from baseline) in the MADRS total score was defined as response criteria. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist (sadness [apparent], sadness [reported], inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts). Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Percentage of participants was calculated by dividing the number of participants meeting response criteria at last visit by the total number of participants analyzed, multiplied by 100%.
Time Frame: Randomization up to 8 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 231 | 221 | 228
percentage of participants | 30.74 | 34.84 | 32.46

8. Secondary Outcome: Change From Randomization to Week 8 in the Hospital Anxiety and Depression Scale (HADS) Depression Subscale Score
Description: as for outcome 6
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 231 | 220 | 228
units on a scale | -3.40 (0.26) | -3.62 (0.27) | -2.55 (0.26)

9. Secondary Outcome: Change From Randomization to Week 8 in Montgomery-Asberg Depression Rating Scale (MADRS) Individual Items
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist (sadness [apparent], sadness [reported], inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts). Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline item score, treatment-by-visit and baseline item score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 231 | 220 | 228
units on a scale
  Apparent sadness | -1.34 (0.08) | -1.25 (0.08) | -1.26 (0.08)
  Reported sadness: number analyzed (Participants) | 231 | 219 | 228
  Reported sadness | -1.41 (0.09) | -1.31 (0.09) | -1.26 (0.09)
  Inner tension | -0.96 (0.08) | -0.91 (0.08) | -0.87 (0.08)
  Reduced sleep | -0.82 (0.09) | -0.96 (0.09) | -0.92 (0.09)
  Reduced appetite | -0.57 (0.08) | -0.67 (0.08) | -0.71 (0.08)
  Concentration difficulties | -1.13 (0.08) | -1.14 (0.08) | -0.98 (0.08)
  Lassitude | -1.15 (0.09) | -1.07 (0.09) | -1.16 (0.09)
  Inability to feel | -1.11 (0.09) | -1.30 (0.09) | -1.14 (0.09)
  Pessimistic thoughts | -0.84 (0.07) | -0.82 (0.07) | -0.91 (0.07)
  Suicidal thoughts | -0.17 (0.03) | -0.19 (0.03) | -0.17 (0.03)

10. Secondary Outcome: Change From Randomization to Week 8 in Clinical Global Impressions of Severity (CGI-S)
Description: CGI-S measures severity of depression at the time of assessment compared with the start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 231 | 220 | 228
units on a scale | -1.20 (0.08) | -1.21 (0.08) | -1.14 (0.07)

11. Secondary Outcome: Change From Randomization to Week 8 in The Fatigue Associated With Depression (FAsD) Average Score and Experience Subscale Score
Description: The FAsD is a participant-rated scale with a total of 13 items. Six of the 13 items ask how often participants experience different aspects of fatigue with responses from 1 (never) to 5 (always). Seven of the 13 items ask how often fatigue impacts various aspects of the participant's lives with responses from 1 (not at all) to 5 (very much). The experience subscale score was derived by taking the mean of Items 1 through 6, and the average score was the mean of Items 1 through 13 (derived by taking the mean of all applicable items for each participant). Item 12 applied only to participants with a spouse or significant other and Item 13 applied to participants who had a job or who went to school. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 225 | 210 | 221
units on a scale
  FAsD average score | -0.67 (0.05) | -0.68 (0.06) | -0.53 (0.05)
  FAsD experience score | -0.63 (0.06) | -0.67 (0.06) | -0.50 (0.06)

12. Secondary Outcome: Change From Randomization to Week 8 in Sheehan Disability Scale (SDS) Items
Description: The SDS was completed by the participant and used to assess the effect of the participant's symptoms on their work (work/school impairment score), social life (social life/leisure activities impairment score), and family life (family life/home responsibilities impairment score). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline item score, treatment-by-visit, and baseline item score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 225 | 210 | 221
units on a scale
  Work impairment score: number analyzed (Participants) | 151 | 138 | 145
  Work impairment score | -1.81 (0.19) | -1.93 (0.20) | -1.32 (0.19)
  Social life impairment score | -1.79 (0.16) | -2.11 (0.16) | -1.52 (0.16)
  Family life impairment score | -1.75 (0.15) | -2.16 (0.15) | -1.47 (0.15)

13. Secondary Outcome: Change From Randomization to Week 8 in the Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF)
Description: The Q-LES-Q-SF is a self-administered 16 item questionnaire measuring degree of enjoyment and satisfaction experienced in various areas of daily life during the past week on a 5-point Likert scale (1=very poor and 5=very good). The total raw score is the sum of Items 1 to 14 and ranges from 14 to 70. The raw scores are converted to and expressed as the percentage of the maximum possible score. Higher scores indicate higher levels of enjoyment/satisfaction. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of maximum possible score
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 224 | 210 | 221
percentage of maximum possible score | 10.54 (1.00) | 10.05 (1.02) | 8.74 (0.99)

14. Secondary Outcome: Change From Randomization to Week 8 in the EuroQol Questionnaire-5 Dimension (EQ-5D)
Description: The EQ-5D Visual Analog Scale is a generic, multidimensional, health-related, quality-of-life instrument. Overall health state score is self-reported using a visual analogue scale, marked on a scale of 0 to 100 with 0 representing worst imaginable health state and 100 representing best imaginable health state. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 225 | 210 | 221
units on a scale | 11.457 (1.218) | 11.895 (1.239) | 9.530 (1.207)

15. Secondary Outcome: Percentage of Participants With Treatment-emergent (TE) Suicidal Ideation and Behaviors Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS captured occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation was defined as a "yes" answer to any 1 of 5 suicidal ideation questions, which included a wish to be dead and 4 different categories of active suicidal ideation. Suicidal behavior was defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation and behavior are defined as treatment-emergent (TE) if not present at baseline. Percentage of participants was calculated by dividing the number of participants with suicide-related TE events by the total number of participants analyzed, multiplied by 100%. A summary of serious and other non-serious adverse events, regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Randomization through 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- 6 mg Fixed Dose LY2216684 + SSRI: LY2216684: fixed dose of 6 mg, administered orally, QD for 8 weeks, adjunctive to an SSRI)
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 232 | 221 | 228
percentage of participants
  TE suicidal ideation | 5.17 | 3.62 | 4.39
  TE suicidal behavior: number analyzed (Participants) | 203 | 198 | 202
  TE suicidal behavior | 0.00 | 0.00 | 0.00

16. Secondary Outcome: Change From Randomization to Week 8 in the Arizona Sexual Experiences (ASEX) Scale
Description: The ASEX scale was used to assess sexual functioning in both males and females. The ASEX total score for the male and female version was calculated as the sum of the responses (rated from 1 [extremely] to 6 [no/never]) of the 5 items of the ASEX scale. Total scores ranged from 5 to 30, with higher scores indicating greater sexual dysfunction. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 224 | 209 | 220
units on a scale | -1.62 (0.29) | -1.29 (0.29) | -0.97 (0.29)

17. Secondary Outcome: Change From Randomization to Week 8 in the Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ)
Description: The CPFQ is a 7-item participant-rated questionnaire pertaining to a participant's cognitive and physical well-being. It assesses motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each item was scored on a 6-point scale ranging from 1 (greater than normal) to 6 (totally absent). Total scores ranged from 7 to 42. Higher scores indicate greater disease severity. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit, and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 225 | 210 | 221
units on a scale | -4.74 (0.38) | -4.67 (0.39) | -3.64 (0.38)

18. Secondary Outcome: Change From Randomization to Week 8 in Blood Pressure
Description: Blood pressure measurements were collected when the participant was in a sitting position. Three measurements of sitting blood pressure collected at approximately 1-minute intervals at every visit were averaged and used as the value for the visit. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline value, treatment-by-visit, and baseline value-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 232 | 220 | 228
millimeters of mercury (mmHg)
  Systolic blood pressure | 1.64 (0.62) | 2.93 (0.63) | 0.78 (0.62)
  Diastolic blood pressure | 3.46 (0.49) | 4.47 (0.50) | 1.01 (0.49)

19. Secondary Outcome: Change From Randomization to Week 8 in Pulse Rate
Description: Pulse measurements were collected when the participant was in a sitting position. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline value, treatment-by-visit, and baseline value-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 12 or 18 mg Flexible Dose LY2216684 + SSRI | 6 mg Fixed Dose LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 232 | 220 | 228
beats per minute (bpm) | 9.26 (0.65) | 7.32 (0.66) | -1.03 (0.65)

20. Secondary Outcome: Pharmacokinetics: Plasma Concentrations of LY2216684
Description: A validated bioanalytical assay was used to determine plasma LY2216684 concentrations.
Time Frame: Pre-randomization, 1 week, 4 weeks, and 8 weeks
Population: Participants exposed to LY2216684 with evaluable plasma concentration values. Samples with concentrations below the lower quantification limit (BQL) of the assay were treated as missing values for the analysis and samples with incomplete dosing information were not included in the pharmacokinetic assessment.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- LY2216684: LY2216684: flexible dose of 12 or 18 milligrams (mg) or fixed dose of 6 mg, administered orally, once daily (QD)
Arm/Group | LY2216684
Number analyzed (Participants) | 400
nanograms per milliliter (ng/mL)
  6-mg dose: number analyzed (Participants) | 197
  6-mg dose | 17.0 (10.2)
  12-mg dose: number analyzed (Participants) | 197
  12-mg dose | 32.2 (21.1)
  18-mg dose: number analyzed (Participants) | 136
  18-mg dose | 52.4 (34.6)

ADVERSE EVENTS:
Groups:
- Placebo + SSRI (Pre-randomized) - CF Phase: Placebo: administered orally, once daily for 3 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Includes all enrolled who did not discontinue for the reason 'Lost to Follow-up' at the first post-baseline visit during the Confirmation (CF) Phase.
- 12 or 18 mg LY2216684 + SSRI (Randomized) - AT Phase: LY2216684: flexible dose of 12 or 18 milligrams (mg), administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Includes randomized participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-randomization visit during the Adjunctive Treatment (AT) Phase.
- 6 mg LY2216684 + SSRI (Randomized) - AT Phase: LY2216684: fixed dose of 6 milligrams (mg), administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Includes randomized participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-randomization visit during the Adjunctive Treatment (AT) Phase.
- Placebo + SSRI (Randomized) - AT Phase: Placebo: administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Includes randomized participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-randomization visit during the Adjunctive Treatment (AT) Phase.
- Placebo + SSRI (Non-randomized) - AT Phase: Placebo: administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Includes all non-randomized participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-randomization visit during the Adjunctive Treatment (AT) Phase.
- Placebo + SSRI (Pre-randomized) - DC Phase: No study drug was administered. Participants were to maintain their selective serotonin reuptake inhibitor (SSRI) treatment at a stable dose for 1 week.
  Includes all enrolled participants who abruptly discontinued placebo after early withdrawal during the Confirmation (CF) Phase and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
- 12 or 18 mg LY2216684 + SSRI (Randomized) - DC Phase; 6 mg LY2216684 + SSRI (Randomized) - DC Phase: No study drug was administered. Participants were to maintain their selective serotonin reuptake inhibitor (SSRI) treatment at a stable dose for 1 week.
  Includes all randomized participants who abruptly discontinued LY2216684 either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
- Placebo + SSRI (Randomized) - DC Phase: No study drug was administered. Participants were to maintain their selective serotonin reuptake inhibitor (SSRI) treatment at a stable dose for 1 week.
  Includes all randomized participants who abruptly discontinued placebo either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
- Placebo + SSRI (Non-randomized) - DC Phase: No study drug was administered. Participants were to maintain their selective serotonin reuptake inhibitor (SSRI) treatment at a stable dose for 1 week.
  Includes all non-randomized participants who abruptly discontinued placebo either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
Arm/Group | Placebo + SSRI (Pre-randomized) - CF Phase | 12 or 18 mg LY2216684 + SSRI (Randomized) - AT Phase | 6 mg LY2216684 + SSRI (Randomized) - AT Phase | Placebo + SSRI (Randomized) - AT Phase | Placebo + SSRI (Non-randomized) - AT Phase | Placebo + SSRI (Pre-randomized) - DC Phase | 12 or 18 mg LY2216684 + SSRI (Randomized) - DC Phase | 6 mg LY2216684 + SSRI (Randomized) - DC Phase | Placebo + SSRI (Randomized) - DC Phase | Placebo + SSRI (Non-randomized) - DC Phase
Serious Adverse Events (participants affected / at risk) | 7/1476 | 2/232 | 1/223 | 2/231 | 5/699 | 3/25 | 0/212 | 2/213 | 1/220 | 2/659
Other Adverse Events (participants affected / at risk) | 231/1476 | 57/232 | 39/223 | 38/231 | 115/699 | 0/25 | 18/212 | 22/213 | 17/220 | 64/659
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo + SSRI (Pre-randomized) - CF Phase (N=1476) | 12 or 18 mg LY2216684 + SSRI (Randomized) - AT Phase (N=232) | 6 mg LY2216684 + SSRI (Randomized) - AT Phase (N=223) | Placebo + SSRI (Randomized) - AT Phase (N=231) | Placebo + SSRI (Non-randomized) - AT Phase (N=699) | Placebo + SSRI (Pre-randomized) - DC Phase (N=25) | 12 or 18 mg LY2216684 + SSRI (Randomized) - DC Phase (N=212) | 6 mg LY2216684 + SSRI (Randomized) - DC Phase (N=213) | Placebo + SSRI (Randomized) - DC Phase (N=220) | Placebo + SSRI (Non-randomized) - DC Phase (N=659)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1/979 (1) | 0/149 (0) | 1/152 (1) | 0/156 (0) | 0/464 (0) | 0/16 (0) | 0/133 (0) | 1/148 (1) | 0/145 (0) | 0/441 (0)
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0/979 (0) | 0/149 (0) | 0/152 (0) | 1/156 (1) | 0/464 (0) | 0/16 (0) | 0/133 (0) | 0/148 (0) | 0/145 (0) | 0/441 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + SSRI (Pre-randomized) - CF Phase (N=1476) | 12 or 18 mg LY2216684 + SSRI (Randomized) - AT Phase (N=232) | 6 mg LY2216684 + SSRI (Randomized) - AT Phase (N=223) | Placebo + SSRI (Randomized) - AT Phase (N=231) | Placebo + SSRI (Non-randomized) - AT Phase (N=699) | Placebo + SSRI (Pre-randomized) - DC Phase (N=25) | 12 or 18 mg LY2216684 + SSRI (Randomized) - DC Phase (N=212) | 6 mg LY2216684 + SSRI (Randomized) - DC Phase (N=213) | Placebo + SSRI (Randomized) - DC Phase (N=220) | Placebo + SSRI (Non-randomized) - DC Phase (N=659)
Tachycardia (Cardiac disorders) | 6 (6) | 12 (12) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 77 (80) | 12 (17) | 12 (13) | 9 (10) | 25 (41) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 13 (13)
Nasopharyngitis (Infections and infestations) | 35 (35) | 12 (12) | 7 (7) | 7 (7) | 27 (27) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 112 (127) | 14 (15) | 15 (18) | 22 (33) | 61 (81) | 0 (0) | 13 (14) | 19 (19) | 14 (14) | 47 (54)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 34 (35) | 18 (19) | 7 (8) | 4 (4) | 11 (11) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days